CLINICAL TRIAL: NCT03306693
Title: Effectiveness of an Educational Intervention Aimed at Increasing the Emotional Competence of Patients With Oesogastric and Bronchopulmonary Cancers as Compared to Standard Management
Brief Title: Educational Intervention to Increase the Emotional Competence of Patients With Oesogastric and Bronchopulmonary Cancers
Acronym: EmoVie_K
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient inclusions
Sponsor: University Hospital, Lille (Other)
Collaborators: SIRIC ONCOLille (Unknown); Santelys Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016_29; 2017-A00224-49 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2017-10-04; First posted 2017-10-11 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Digestive System Neoplasms; Thoracic Neoplasms
Keywords: Emotional Intelligence; Quality of Life
MeSH Terms: conditions — Digestive System Neoplasms; Thoracic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emotional skills (Experimental): 3 group sessions where patients are going to learn how to identify, express and regulate their emotions
  Interventions: Behavioral: Emotional skills
- Relaxation and talking group (Sham Comparator): 3 group sessions where patients are going to follow relaxation instructions and after a non directive talking group about cancer
  Interventions: Behavioral: Relaxation and talking group

INTERVENTIONS:
Behavioral: Emotional skills — 2-hour 3 group sessions
  Other Names: Emotional intelligence
  Arms: Emotional skills
Behavioral: Relaxation and talking group — 2-hour 3 group sessions
  Arms: Relaxation and talking group

SUMMARY:
The aim of this study is to test whether a short educational intervention about emotional skills can improve survivor cancer patient emotional skills and quality of life. Half of participants will follow the educational intervention about emotional skills, while the other half will practice relaxation followed by a non-directive talking group. The educational intervention should give better results on patient emotional skills and quality of life than the control group.

DETAILED DESCRIPTION:
After the end of treatments, cancer patients face a difficult time because it is expected that they return to normal, but at the same time they still have to struggle with the aftermath of cancer and fear of recurrence. This is why there is room in this period for an intervention designed to help patients to cope with their emotions. . Patient emotional skills are patient abilities to identify, express and manage their emotions for the best possible psychological adjustment. In general population, emotional skills have been shown to be highly related to a better quality of life. In this randomized controlled study, bronchopulmonary and oesogastric cancer patients between 6 months and 2 years after the end of treatments will undergo either the emotional skills intervention (intervention group) or the relaxation group (control group).

ELIGIBILITY:
Inclusion Criteria:

* ≥18 ans,
* Oesogastric or bronchopulmonary cancer patients between 6 months and 2 years after the end of cancer treatments
* Patient of the CHRU (Regional Teaching Hospital) of Lille,
* Registered with a social security scheme
* Speak and understand French language
* Signature of the informed consent to participate in the study.

Exclusion Criteria:

* Cognitive disorders or unstabilized psychiatric disorders that may impair the ability of reasoning and thinking necessary to complete the questionnaires and attend workshops
* Difficulty or deficiency that prevent the patient from a good understanding of the imperatives of the research
* Any situation likely to significantly affect emotional competence during the study according to the investigator's judgment (in particular, ongoing psychotherapy )
* Patients under judicial protection (guardianship or curators).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2019-05-07 (Actual); Study Completion 2019-05-07 (Actual)

PRIMARY OUTCOMES:
Change in patient emotional skills from baseline to 15 days after intervention | Baseline and 15 days after the end of the intervention
  Variation of patient-reported Short Profile of Emotional Competence (S-PEC)questionnaire score from baseline to 15 days after the intervention (between 1 and 3 months)

SECONDARY OUTCOMES:
Patient emotional skills long term | T1 (15 days after the end of the intervention) and T2 (2 months after T1) : 2 months
  Variation of patient-reported PEC (Profile of Emotional Competence) questionnaire score
Quality of life by Medical Outcome Study Health Survey Short Form-36 (MOS SF-36) | Baseline (T0), 15 days after the end of the intervention (T1), 2 months
  Patient-reported health-related quality of life using the Medical Outcome Study Health Survey Short Form-36 (MOS SF-36)
Patient participation in workshops | Between 2 weeks and 2 months
  The percentage of patients who have attended the 3 group sessions
Patient adherence to exercises to do at home between sessions | Between 2 weeks and 2 months
  The percentage of patients who have performed the suggested exercises at home between sessions
Patient satisfaction | T1 (15 days after the end of the intervention) and T2 (2 months after T1)
  Patient-reported satisfaction regarding the intervention using and ad hoc questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Calmette,CHU, Lille, France